CLINICAL TRIAL: NCT03699813
Title: Use of Rotational Thromboelastometry (ROTEM) in Pediatric Perioperative Medicine and Its Comparison With Standard Coagulation Tests aPTT/PT
Brief Title: ROTEM Versus aPTT/PT in Pediatric Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Durila Miroslav MUDr. Ph.D., associated professor, University Hospital, Motol
Other Study IDs: 05102018
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Coagulation Defect; Bleeding
Keywords: ROTEM, PT, aPTT
MeSH Terms: conditions — Hemostatic Disorders; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- scoliosis bleeding management based on aPTT/PT: Bleeding and coagulopathy during surgery managed by clinical approach and aPTT/PT tests.
  Blood loss, consumption of fresh frozen plasma (FFP), red blood cell units consumption and time to aPTT/PT tests result will be analysed.
  Interventions: Other: Comparison of two approaches to bleeding management
- scoliosis bleeding management based on ROTEM: Bleeding and coagulopathy during surgery managed by ROTEM. Blood loss, consumption of fresh frozen plasma (FFP), red blood cell units consumption and time to aPTT/PT tests result will be analysed.
  Interventions: Other: Comparison of two approaches to bleeding management

INTERVENTIONS:
Other: Comparison of two approaches to bleeding management

SUMMARY:
Hemocoagulation management in perioperative bleeding is nowadays based on standard coagulation testing: activated partial thromboplastin time (aPTT), prothrombin time (PT), fibrinogen, D-dimers, platelets. An interest about viscoelastic coagulation testing methods is rising - use of rotational thromboelastometry (ROTEM) is mentioned in the newest European guidelines for hemostasis management. ROTEM has more advantages then standard tests. However, both tests have only grade 1C recommendation, and most of trials have been done on adults. The goal of the study is to compare a relationship between standard tests and ROTEM in pediatric patients in perioperative period to find out which test has better correlation with clinical status, to compare therapeutic strategies and time necessary for gain both of tests and to compare the difference in blood loss and blood products consumption in group treated by ROTEM versus standard tests. Reduced blood loss and amount of blood products transfusion is expected to be found in ROTEM group, representing lowering risk for the patient, all due to early evaluation of hemocoagulation and targeted therapy guided by ROTEM.

DETAILED DESCRIPTION:
Pediatric patients who underwent spine surgery (under 18 years old) will be recruited in our study.

Retrospective data will be analysed from these patient who underwent scoliosis surgery before ROTEM implementation to daily practice and after ROTEM implementation do daily practice in our department.

Time to available results of ROTEM versus aPTT/PT tests will be compared. Blood loss and blood products used in these both groups will be analysed and compared between 2 groups.

ELIGIBILITY:
Inclusion Criteria:

• pediatric patients after surgical correction of scoliosis

Exclusion Criteria:

• patients older than 18 years

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients who underwent surgical scoliosis correction
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
analysing blood loss during surgery | 3 years
  blood loss during scoliosis surgery will analysed in both groups

SECONDARY OUTCOMES:
analysing blood transfusion units consumption | 3 years
  consumption of blood transfusion products will be analysed in both groups
time to results of tests | 3 years
  time to available results of test ROTEM and aPTT/PT will be analysed and compared between both groups

IPD SHARING:
Plan to Share IPD: Undecided
All data of study will be available in published paper

REFERENCES:
- [Derived] Jonas J, Durila M, Malosek M, Maresova D, Stulik J, Barna M, Vymazal T. Usefulness of perioperative rotational thrombelastometry during scoliosis surgery in children. J Neurosurg Spine. 2020 Jan 24;32(6):865-870. doi: 10.3171/2019.11.SPINE191137. Print 2020 Jun 1. PMID 31978886